CLINICAL TRIAL: NCT00810563
Title: Assessment of Postoperatory Pain After Laparoscopic Tubal Ligation by Electrocoagulation With Bupivacaine or Placebo
Brief Title: Does Bupivacaine in Laparoscopic Portals Reduce Post Surgery Pain in Tubal Ligation by Electrocoagulation?
Acronym: DOPOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Ricardo Francalacci Savaris, HCPA - UFRGS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DOPOL 08-294; GPPG 08-293
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Pain
Keywords: pain; tubal ligation; bupivacaine; laparoscopy
MeSH Terms: conditions — Pain | interventions — Saline Solution; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Saline solution 0.9% 5mL in each portal
  Interventions: Drug: Saline solution (laparoscopic tubal ligation)
- 2 (Active Comparator): Bupivacaine 0.5% 5mL in each portal
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Saline solution (laparoscopic tubal ligation) — 5ml of saline solution in each portal of the trocar (2 portals)
  Arms: 1
Drug: Bupivacaine — 5ml of bupivacaine 0.5% in each trocar portal
  Arms: 2

SUMMARY:
The use of bupivacaine , an anesthesic, in laparoscopic portals is recommended in some surgeries. In the ase of tubal ligation by electrocoagulation, where pain is reduced, there is no evidence of this benefit. The objective of this study is to verify the degree of pain after laparoscopic tubal ligation surgery in patient who received bupivacaine 0.5% in the portal, or placebo

DETAILED DESCRIPTION:
In order to conduct this study, the internal and external validation were considered.

The author will use different gynecological teams, with different expertise to perform the laparoscopic tubal ligation, but using the same surgical and anesthesic technique. Second year residents, during their rotation, and medical staff will perform the surgery.

Anesthesic technique:

Intravenous remifentanil 0.1-0.5 micrograms/kg/min Intravenous Propofol target controlled or sevoflurane Intermittent ventilation using O2 40 - 100%, with or without compressed air. Before incision: 5mL of bupivacaine 0.5% or saline solution 0.9% from the aponeurosis until the skin In the end of the procedure: intravenous 4mg of dexamethasone + 40mg of tenoxican

Post-operation prescription:

NPO util well awake, then free according to patient´s tolerance If nausea/vomit: metoclopramide 10mg IV If pain: dipyrone 1g IV qid If pain is intense: morphine 3mg IV 3/3 h If pain persists: morphine 1mg h/h

After hospital discharge:

If pain: sodium diclofenac 50mg tid

ELIGIBILITY:
Inclusion Criteria:

* All patients schedule for laparoscopic tubal ligation

Exclusion Criteria:

* Not willing to consent
* Use of analgesic within 12 hours prior the surgery
* Known allergy or contraindications to bupivacaine, dipyrone, porphine, or sodium diclofenac

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-03 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Pain | at 15, 30 and 120 minutes and 14 hours after surgery

SECONDARY OUTCOMES:
Use of medication for pain | at 15, 30 and 120 minutes after surgery and 14 hours later

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Savaris, MD, Principal Investigator — HCPA/UFRGS
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Rioux JE, Daris M. Female sterilization: an update. Curr Opin Obstet Gynecol. 2001 Aug;13(4):377-81. doi: 10.1097/00001703-200108000-00002. PMID 11452199
- [Background] Alexander JI. Pain after laparoscopy. Br J Anaesth. 1997 Sep;79(3):369-78. doi: 10.1093/bja/79.3.369. No abstract available. PMID 9389858
- [Background] Colbert ST, Moran K, O'Hanlon DM, Chambers F, Moriarty DC, Blunnie WP. An assessment of the value of intraperitoneal meperidine for analgesia postlaparoscopic tubal ligation. Anesth Analg. 2000 Sep;91(3):667-70. doi: 10.1097/00000539-200009000-00032. PMID 10960397
- [Background] Curry CS, Darby JR, Janssen BR. Evaluation of pain following electrocautery tubal ligation and effect of intraoperative fentanyl. J Clin Anesth. 1996 May;8(3):216-9. doi: 10.1016/0952-8180(95)00233-2. PMID 8703457
- [Background] Chi IC, Cole LP. Incidence of pain among women undergoing laparoscopic sterilization by electrocoagulation, the spring-loaded clip, and the tubal ring. Am J Obstet Gynecol. 1979 Oct 1;135(3):397-401. doi: 10.1016/0002-9378(79)90713-0. PMID 158312
- [Derived] Savaris RF, Chicar LL, Cristovam RS, Moraes GS, Miguel OA. Does bupivacaine in laparoscopic ports reduce postsurgery pain in tubal ligation by electrocoagulation? A randomized controlled trial. Contraception. 2010 Jun;81(6):542-6. doi: 10.1016/j.contraception.2009.12.019. Epub 2010 Feb 10. PMID 20472124